CLINICAL TRIAL: NCT03707431
Title: A Randomized Trial of a Web-based Non-pharmacological Pain Intervention for Pediatric Chronic Pancreatitis
Brief Title: Internet Based Cognitive Behavioral Therapy in Pediatric Chronic Pancreatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: University of Iowa (Other); University of Virginia (Other); Washington University School of Medicine (Other); M.D. Anderson Cancer Center (Other); The University of Texas Health Science Center, Houston (Other); Children's Hospital Medical Center, Cincinnati (Other); Children's Hospital Los Angeles (Other); Children's Hospital of Philadelphia (Other); University of Toronto (Other); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); Medical College of Wisconsin (Other); Massachusetts General Hospital (Other); University of Minnesota (Other); Ohio State University (Other); University of Pittsburgh (Other); University of California, San Francisco (Other); University of Utah (Other); Indiana University (Other); Sydney Children's Hospitals Network (Other); Cedars-Sinai Medical Center (Other); Stanford University (Other); Ariel Precision Medicine (Industry); University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Tonya Palermo, Professor, Anesthesiology and Pain Medicine, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1R01DK118752-01 (NIH)
Record Dates: First submitted 2018-10-02; First posted 2018-10-16 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Chronic Pancreatitis; Acute Recurrent Pancreatitis
Keywords: Adolescent; Pancreatitis; Pain; Internet Intervention; Behavioral Intervention
MeSH Terms: conditions — Pancreatitis, Chronic; Pancreatitis; Pain

STUDY DESIGN:
Intervention Model Description: Randomized and double-blinded controlled trial of web-based CBT (WebMAP) vs pain education (WebED).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Web-based CBT (WebMAP) (Experimental): Receives access to WebMAP
  Interventions: Behavioral: Web-based CBT
- Pain Education (WebED) (Active Comparator): Receives access to WebED
  Interventions: Behavioral: Pain Education

INTERVENTIONS:
Behavioral: Web-based CBT — The eight child modules include: 1) education about chronic pain, 2) recognizing stress and negative emotions, 3) deep breathing and relaxation, 4) implementing coping skills at school, 5) cognitive skills (e.g., reducing negative thoughts), 6) lifestyle interventions, 7) staying active (e.g., pleasant activity scheduling), 8) relapse prevention. The eight parent modules are: 1) education about chronic pain, 2) recognizing stress and negative emotions, 3) operant strategies I (using attention and praise to increase coping), 4) operant strategies II (using rewards to increase positive coping and reach school goals), 5) modeling, 6) lifestyle, 7) communication, 8) relapse prevention.
  Other Names: WebMAP
  Arms: Web-based CBT (WebMAP)
Behavioral: Pain Education — The pain education website provides publicly available educational information about pancreatitis and abdominal pain. There is general information about pancreatitis from available web sources (e.g., National Pancreas Foundation) as well as information about chronic pain in childhood. The content does not include any instruction in the behavioral and cognitive skills taught within the WebMAP program.
  Other Names: WebED
  Arms: Pain Education (WebED)

SUMMARY:
Abdominal pain is common in children with chronic and acute recurring pancreatitis (CP, ARP), and as they continue into adulthood, the disease progresses with increased pain and greater exposure to opioids. Despite the relevancy of early pain self-management for childhood pancreatitis, there have been no studies of non-pharmacological pain intervention in this population. The proposed project will evaluate a web-based cognitive behavioral pain management program delivered to a cohort of well-phenotyped children with CP/ARP and some community participants to reduce pain, pain-related disability and enhance HRQOL; it will also identify genetic risk factors and clinical and behavioral phenotypic factors associated with treatment response to enable precision medicine approaches.

DETAILED DESCRIPTION:
Abdominal pain is present in 81% of children and adolescents with CP and ARP. Effective treatments that target pain in these children will lessen the risk of opioid exposure and continued pain and disability into adulthood. We plan to recruit a large multicenter sample of 260 children and adolescents (ages 10-19 years) with CP/ARP and their parents from INSPPIRE 2 (INSPPIRE:INternational Study Group of Pediatric Pancreatitis: In search for a cuRE) centers and pancreatitis community groups (e.g. NPF) to evaluate the efficacy of WebMAP, a web-based cognitive behavioral pain management program (CBT). The study design is a two (group) x three (time point) randomized, controlled, double-blinded trial. Participants will be randomly assigned to receive online access to either pain education (WebED) or CBT (WebMAP) over an 8-10 week treatment period. The primary study outcome is abdominal pain symptoms measured at pre-treatment, immediately post-treatment, and at 6-month follow-up. Secondary outcomes include pain-related disability, health-related quality of life, depression and anxiety symptoms, and medication use. This project represents a significant advance in pain management for children with CP/ARP by evaluating the first ever nonpharmacologic pain intervention in these patients, which may guide future developments in the management of chronic pain associated with CP/ARP.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with CP or ARP
2. ages 10-19 years
3. at least 4 acute pancreatitis flare-ups/attacks in past year, or at least 1 instance of moderate (4/10 pain) pancreatitis/abdominal pain in the past month
4. access to the Internet on any web-enabled device

Exclusion criteria:

1. non-English speaking
2. inability to read at the 5th grade level due to learning problem or developmental delay
3. children with cystic fibrosis who have pancreatic insufficiency at the time of diagnosis
4. patients with Shwachman-Bodian-Diamond Syndrome
5. Acute Recurrent Pancreatitis (ARP) with no evidence of chronic or persistent pain
6. anticipated surgery (TPIAT or other) during study participation

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Change in abdominal pain severity | Baseline, 12 weeks, 6 months
  The Abdominal Pain Index (API) assesses characteristics of abdominal pain during the previous 2 weeks including the number of days with pain, number of pain episodes per day, typical pain episode duration, and typical pain intensity. An index is computed with higher scores indicating greater abdominal pain severity.

SECONDARY OUTCOMES:
Change in pain-related disability | Baseline, 12 weeks, 6 months
  The Child Activity Limitations Interview (CALI-9) is a daily diary validated to assess perceived difficulty in completing 9 daily activities as a measure of pain-related disability. Responses are rated on a 5-point scale (0-4) with higher scores indicating greater perceived difficulty with activities. Youth will provide ratings daily for 7 days on their online diaries at each assessment period. Mean total activity limitations across the reporting period is used in analyses, with higher scores indicating greater disability.
Change in health-related quality of life | Baseline, 12 weeks, 6 months
  The Pediatric Quality of Life Inventory (Peds-QL) assesses several domains of functioning, including physical, social, emotional, and academic functioning. The PedsQL is widely used as it demonstrates good reliability for both the parent and child self-report measures. Higher scores indicate fewer difficulties (better) health-related quality of life. Sub scales of physical and psychosocial health will be used in analyses.
Change in emotional distress | Baseline, 12 weeks, 6 months
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Emotional Distress Scales include an 8-item scale of anxiety that assesses fear (e.g., fearfulness), anxious misery (e.g., worry) and hyperarousal (e.g., nervousness) and 8-item scale of depressive symptoms that evaluates negative mood, view of self and social cognitions. Raw scores and T-scores are computed with T-scores above 60 indicating clinically elevated symptoms.
Change in opioid use | Baseline, 12 weeks, 6 months
  Youth and parents will report on over the counter and prescription (opioid and non-opioid) medication use in the preceding 7 days.
Change in pain self-efficacy | Baseline, 12 weeks, 6 months
  The Pain Self-Efficacy Scale is a 7-item measure that assesses the child's beliefs in carrying out activities when in pain. The scale has demonstrated good internal consistency, cross-informant reliability with parent report, and strong construct validity. Higher scores indicate higher self-efficacy.
Change in parent impact of pain | Baseline, 12 weeks, 6 months
  Parents will complete the Bath Adolescent Pain Questionnaire-Parent Impact Questionnaire (BAPQ-PIQ), a measure of the impact of parenting an adolescent with chronic pain. The BAPQ-PIQ is a 62-item questionnaire with 8 scales including: depressive symptoms, anxiety, pain catastrophizing, self-blame, partner relationship, social functioning, parental behavior, and parental role strain. Items are rated on a 5-point frequency response scale (0 = never, 4 = always) with higher scores indicating more impaired functioning for all subscales. The BAPQ-PIQ has demonstrated good reliability and validity among parents of youth with chronic pain. Sub scales will be analyzed separately.
Change in pain interference | Baseline, 12 weeks, 6 months
  The PROMIS Pain Interference - Pediatric Short Form includes 8 items to assess consequences of pain on relevant aspects of one's life. This includes the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities. The scale has been validated in pediatric patients with chronic pain. Raw scores and T-scores are computed with T-scores above 60 indicating clinically elevated symptoms.
Change in health service utilization | Baseline, 6 months
  Parents will complete the Client Service Receipt Inventory-Pain version, a measure of service use, out-of-pocket expenses, and lost work time incurred by families for the evaluation or management of the child's chronic pain. Questions pertain to hospital admissions, outpatient services, community services (e.g., tutor, lawyer), medications, lost work time, paid help, and other costs. We will compute the following variables: total number of services used by category, number of lost parental work days, and number of out-of-pocket expenses.
  visits, medications, other treatments, and indirect costs as reported by the parent.

CONTACTS AND LOCATIONS:
Overall Officials: Tonya Palermo, PhD, Principal Investigator — Seattle Children's Hospital; Aliye Uc, MD, Principal Investigator — University of Iowa
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

REFERENCES:
- [Background] Palermo TM, Murray C, Aalfs H, Abu-El-Haija M, Barth B, Bellin MD, Ellery K, Fishman DS, Gariepy CE, Giefer MJ, Goday P, Gonska T, Heyman MB, Husain SZ, Lin TK, Liu QY, Mascarenhas MR, Maqbool A, McFerron B, Morinville VD, Nathan JD, Ooi CY, Perito ER, Pohl JF, Schwarzenberg SJ, Sellers ZM, Serrano J, Shah U, Troendle D, Zheng Y, Yuan Y, Lowe M, Uc A; Consortium for the Study of Chronic Pancreatitis, Diabetes and Pancreatic Cancer. Web-based cognitive-behavioral intervention for pain in pediatric acute recurrent and chronic pancreatitis: Protocol of a multicenter randomized controlled trial from the study of chronic pancreatitis, diabetes and pancreatic cancer (CPDPC). Contemp Clin Trials. 2020 Jan;88:105898. doi: 10.1016/j.cct.2019.105898. Epub 2019 Nov 19. PMID 31756383